CLINICAL TRIAL: NCT00061152
Title: An Open-Label Pilot Study of High-Concentration Capsaicin Patches in the Treatment of Painful HIV-Associated Neuropathy
Brief Title: Pilot Study of High-Concentration Capsaicin Patches in the Treatment of Painful HIV-Associated Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeurogesX (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: C109
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: Pain Measurement; Diary; Painful HIV Neuropathy; HIV Neuropathy; Capsaicin; Analgesics/*therapeutic use; Capsaicin/*administration & dosage/adverse effects; Peripheral Nervous System Diseases/*complications/diagnosis/*therapy; Peripheral Nervous System Diseases/drug therapy/*etiology/physiopathology; Pain
MeSH Terms: conditions — HIV Infections; Pain

INTERVENTIONS:
Drug: Capsaicin Dermal Patch

SUMMARY:
The purpose of the study is to gain initial information on the tolerability and feasibility of high-concentration capsaicin patches for the treatment of painful HIV-associated neuropathy, whether resulting from HIV disease and/or antiretroviral drug exposure. The study will also provide preliminary safety and efficacy information.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age.
* Documented evidence of HIV-1 infection.
* Painful HIV-associated neuropathy, whether resulting from HIV disease and/or antiretroviral drug exposure, with primary symptoms of pain, burning or dysesthetic discomfort in both feet for at least 2 months prior to Screening Visit.

AND:

* Diminished ankle reflexes (compared to the knee) or absent ankle reflexes,

AND/OR

* Distal diminution of either vibration sensation or pain or temperature sensation in the legs.
* Either no neurotoxic antiretroviral (i.e., didanosine [ddI], zalcitabine [ddC], or stavudine [d4T]) exposure for at least 8 weeks prior to Screening Visit,

OR

* Currently on stable dose(s) of any of the neurotoxic antiretrovirals listed above for at least 8 weeks prior to Screening Visit, without a foreseeable need to change doses or medications for duration of study.
* Screening Pain Sum Score of 12 to 36.
* Intact, unbroken skin over the painful area(s) to be treated.
* If taking chronic pain medications, be on a stable (not PRN) regimen for at least 7 days prior to Treatment Visit (Day 0) and willing to maintain medications at same stable dose(s) and schedule throughout the study.
* Be willing and able to use Roxicodone® (oxycodone) oral solution, if needed, to relieve treatment-associated discomfort.
* Female subjects with child-bearing potential must have a negative urine or serum pregnancy test, to be performed at the Screening Visit.
* All subjects must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study and for 30 days following experimental drug exposure.
* Be willing and able to comply with protocol requirements for the duration of study participation. (Such requirements include, but are not limited to: completing a daily pain diary, attending all study visits, and refraining from extensive travel during study participation.)

Exclusion Criteria:

* Presence of acute, active opportunistic infection, except oral thrush; oral, genital, or rectal herpes; and Mycobacterium avium bacteremia within 2 weeks prior to Screening Visit.
* Significant pain of an etiology other than painful HIV-associated neuropathy, for example, compression-related neuropathies, e.g., spinal stenosis, or fibromyalgia or arthritis. Subjects must not have significant ongoing pain from other cause(s) that may interfere with judging HIV-associated neuropathy pain.
* Evidence of another contributing cause for peripheral neuropathy, e.g., diabetes mellitus, hereditary neuropathy, vitamin B12 deficiency (B12 level less than or equal to 200 pg/mL) or less than 3 months of B12 supplementation prior to Screening Visit, or treatment within 90 days prior to Screening Visit with any drug that may have contributed to the sensory neuropathy.
* Any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain.
* Recent use (within 21 days preceding the Treatment Visit [Day 0]) of any topically applied pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics (including Lidoderm®), steroids or capsaicin products on the painful areas.
* Treatment for acute opportunistic infections within 14 days before Treatment Visit (Day 0). Maintenance treatment of cytomegalovirus (CMV) retinitis, Mycobacterium avium bacteremia, or cryptococcal meningitis is permitted.
* Current use of any investigational drug, or Class 1 anti-arrhythmic drugs (such as tocainide and mexiletine).
* Hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics, Roxicodone or adhesives.
* Significant ongoing or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function that may interfere either with the ability to complete the study or the evaluation of adverse events.
* Currently have active malignant disease. Malignancies in remission that do not require further treatment or Kaposi's sarcoma requiring local treatment only are allowed.
* High tolerance to opioids that precludes the ability to relieve treatment-associated discomfort with Roxicodone® if needed, as judged by investigator.
* History or current problem with prescription drug, illicit substance, or alcohol abuse from self report or as judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - NeurogesX Investigational Site, West Hollywood, California
  - NeurogesX Investigational Site, New York, New York
  - NeurogesX Investigational Site, Portland, Oregon